CLINICAL TRIAL: NCT03614364
Title: Combination of Nanoxel and Herzuma as First-line Chemotherapy in Patients With Metastatic Salivary Duct Carcinoma : Open Label Single Arm Multicenter Phase II Study
Brief Title: Combination of Nanoxel and Herzuma in Salivary Duct Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-11-082
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Salivary Duct Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nanoxel and herzuma (Experimental): D1 Nanoxel 75 mg/m2 + D5W 100mL MIV over 1hr D1 Herzuma 8mg/kg (loading dose) + N/S 250mL miv over 90mins 6mg/kg (maintenance) + N/S 250mL MIV over 30mins (since 2 cycle) repeated every 3 weeks
  Interventions: Drug: nanoxel; Drug: herzuma

INTERVENTIONS:
Drug: nanoxel — D1 Nanoxel 75 mg/m2 + D5W 100mL MIV over 1hr D1 Herzuma 8mg/kg (loading dose) + N/S 250mL miv over 90mins 6mg/kg (maintenance) + N/S 250mL MIV over 30mins (since 2 cycle) repeated every 3 weeks
Drug: herzuma — D1 Nanoxel 75 mg/m2 + D5W 100mL MIV over 1hr D1 Herzuma 8mg/kg (loading dose) + N/S 250mL miv over 90mins 6mg/kg (maintenance) + N/S 250mL MIV over 30mins (since 2 cycle) repeated every 3 weeks

SUMMARY:
1. Study outline This is a multicenter, single-arm, phase II trial to evaluate the efficacy and safety of nanoxel plus herzuma combination chemotherapy in patients with metastatic salivary ductal cancer. Approximately 41 patients will be enrolled. Treatment will be continued until disease progression or unacceptable toxicities. Response evaluation will be performed every 2 cycles.
2. Dosing & Treatment schedule D1 Nanoxel 75 mg/m2 + D5W 100mL MIV over 1hr D1 Herzuma 8mg/kg (loading dose) + N/S 250mL miv over 90mins 6mg/kg (maintenance) + N/S 250mL MIV over 30mins (since 2 cycle) repeated every 3 weeks (In case of discontinuation of nanoxel without progression, single agent herzuma can be administered until progression)

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed HER2 positive (immunohistochemistry [IHC] 3+, and/or fluorescence in situ hybridization[FISH] positive with ≥ two-fold amplification) salivary duct carcinoma(SDC), and other salivary gland carcinomas which are similar to SDC in histopathological findings, including adenocarcinoma, not otherwise specified, acinic cell carcinoma, squamous cell carcinoma, anaplastic carcinoma, high grade mucoepidermoid carcinoma, and carcinoma ex pleomorphic adenoma
* stage IV or recurrent cancer
* age ≥ 20 years
* ECOG performance status 0-2
* At least one measurable tumor lesion according to RECIST 1.1
* Expected survival for approximately 12 weeks or longer
* No prior systemic chemotherapy
* At least 4 weeks later after surgery or radiotherapy
* Written informed consent

Exclusion Criteria:

* Severe or unstable cardiac disease, including (for example) coronary artery disease requiring increased doses of anti-anginal medication and/or coronary angioplasty (including stent placement) within the preceding 24 months(congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias)
* Uncontrolled systemic illness such as DM, hypertension, hypothyroidism and infection
* Pregnant and nursing women (women of reproductive potential have to agree to use an effective contraceptive method)
* Current, known CNS malignancy (history of completely resected or irradiated brain metastases by WBRT or stereotactic radiosurgery allowed)
* Patients with alcohol abuse

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Response rate | about 24months
  according to RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided